CLINICAL TRIAL: NCT00213447
Title: Characterization of T Cell Response in Hypersensitivity Syndrome
Brief Title: T Cell Response in Hypersensitivity Syndrome
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2001/056/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Hypersensitivity; Syndrome
MeSH Terms: conditions — Hypersensitivity; Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
immunological study of the T cell repertoire phenotype and functionality in hypersensitivity syndrome.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* cutaneous eruption
* lymph nodes
* hepatitis
* interstitial pneumonia
* nephritis
* cardiopathy
* eosinophilia
* hyperlymphocytosis

Exclusion Criteria:

* age minor to 18
* HIV +

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Drug rash with eosinophilia and systemic symptoms
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2002-11; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Joly, MD-PHD, Principal Investigator — UH rouen
Locations (1):
- UH-Rouen, Rouen, France

REFERENCES:
- [Derived] Picard D, Janela B, Descamps V, D'Incan M, Courville P, Jacquot S, Rogez S, Mardivirin L, Moins-Teisserenc H, Toubert A, Benichou J, Joly P, Musette P. Drug reaction with eosinophilia and systemic symptoms (DRESS): a multiorgan antiviral T cell response. Sci Transl Med. 2010 Aug 25;2(46):46ra62. doi: 10.1126/scitranslmed.3001116. PMID 20739682